CLINICAL TRIAL: NCT06905236
Title: Kidney Function Markers in Postmenopausal Obese Women: Response to Aerobic Training
Brief Title: Kidney Function in Obese Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wissal Abassi (Other)
Responsible Party: Sponsor-Investigator, Wissal Abassi, Principal Investigator, High Institute of Sports and Physical Education of Kef
Organization: High Institute of Sports and Physical Education of Kef (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Training and kidney
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Kidney Function Tests
Keywords: Glomerular Filtration Rate; neutrophils; obesity; serum creatinine; walking training; white blood cells
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training group (Experimental): The training group underwent a moderate intensity intermittent walking training at 60% to 80% of the 6- min-walking-test distance, four times a week of 60 min/session for a period of 10 weeks.
  Interventions: Behavioral: walking intervention
- Control group (No Intervention): No training intervention was intended for the control group.

INTERVENTIONS:
Behavioral: walking intervention — Moderate intensity intermittent walking training for a period of 10 weeks. The intensity of the training is 60 to 80% of 6MWTdistance. The frequency of the training is four times a week.
  Arms: Training group

SUMMARY:
The goal of this clinical trial is to investigate the impact of a 10-week moderate intensity interval walking training (MIIWT) program on kidney function markers in obese postmenopausal women. The main question it aims to answer is:

Does MIIWT improve kidney function markers in this population? Researchers will compare MIIWT (designed to training group) to non-training intervention (designed to control group) to see if the training program works to improve kidney function markers.

Participants in training group will: perform a 10-week MIIWT program, four sessions per week (5 repetitions of 6-min-walking-test (6MWT) at 60-80% of 6MWTdistance measured at baseline, interspersed by 6-min of active recovery between repetitions). Participants in control group will : not perform any physical training and maintain their usual daily activities.

DETAILED DESCRIPTION:
The convergence of the obesity pandemic and the postmenopausal status is likely associated with renal function decline. Regular aerobic training have been shown to prevent adverse health outcomes in obese. The main purpose of this study was to evaluate changes in kidney function markers and white blood cell (WBC) subpopulations in obese postmenopausal women participating in moderate intensity interval walking training (MIIWT). A total of 36 obese postmenopausal women were randomized to MIIWT (CON, n=18) or control group (CON, n=18), four times a week for 10-week. The MIIWT consisted on 5 repetitions of walking for 6-min at 60-80% of the 6-min-walk-test-distance with 6-min of active recovery between repetitions. Before and after the MIIWT, body composition, kidney function markers (serum creatinine [sCr], blood urea nitrogen [BUN], serum uric acid [sUA] and Glomerular Filtration Rate [GFR] and white blood cells (WBC) count and its specific subpopulations (neutrophils [NEU], lymphocytes [LYM], monocytes [MON], eosinophils [EOSI] and basophils [BASO]) were assessed.

ELIGIBILITY:
Inclusion Criteria:

* be aged between 50 and 60 years.
* be postmenopausal (absence of menses > 12 months).
* present a BMI greater than or equal to 30 kg/m2.
* be free of any special diets in the three months prior to the start of the intervention.
* have a sedentary lifestyle (exercise less than 2 h/week).

Exclusion Criteria:

* Suffering from any cardiovascular/renal/pulmonary/metabolic disease.
* Being under menopausal hormone therapy.
* Presenting any orthopedic limitations interfering the ability to perform the study intervention.

Ages: 50 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2024-09-23 (Actual); Primary Completion 2024-12-22 (Actual); Study Completion 2024-12-22 (Actual)

PRIMARY OUTCOMES:
serum creatinine | At baseline and at week 11(after the ten weeks of the training intervention).
  serum concentrations of creatinine (sCr) are measured from a blood sample (5 ml) using a Chemistry System Analyzer (Beckman Coulter AU480, France).
blood urea nitrogen | At baseline and at week 11(after the ten weeks of the training intervention).
  serum concentrations of blood urea nitrogen (BUN) are measured from a blood sample (5 ml) using a Chemistry System Analyzer (Beckman Coulter AU480, France).
serum uric acid | At baseline and at week 11(after the ten weeks of the training intervention).
  serum concentrations of uric acid (sUA) are measured from a blood sample (5 ml) using a Chemistry System Analyzer (Beckman Coulter AU480, France).
glomerular Filtration Rate | At baseline and at week 11(after the ten weeks of the training intervention).
  the glomerular Filtration Rate (GFR) has been computed using the Cockcroft formula, as follows: GFR (mL/min) = [(140 - age) × weight ×0.85]/(sCr× 72).
white blood cells count | At baseline and at week 11(after the ten weeks of the training intervention).
  blood concentration of white blood cells (WBC) count were collected (5 ml) in test tubes containing EDTA and analyzed using an automated cell counter (XN450; Sysmex, Norderstedt, Germany)
neutrophils | At baseline and at week 11(after the ten weeks of the training intervention).
  blood concentration of neutrophils (NEU) were collected (5 ml) in test tubes containing EDTA and analyzed using an automated cell counter (XN450; Sysmex, Norderstedt, Germany).
lymphocytes | At baseline and at week 11(after the ten weeks of the training intervention).
  blood concentrations of lymphocytes (LYM) were collected (5 ml) in test tubes containing EDTA and analyzed using an automated cell counter (XN450; Sysmex, Norderstedt, Germany).
monocytes | At baseline and at week 11(after the ten weeks of the training intervention).
  blood concentration of monocytes (MON) were collected (5 ml) in test tubes containing EDTA and analyzed using an automated cell counter (XN450; Sysmex, Norderstedt, Germany).
eosinophils | At baseline and at week 11(after the ten weeks of the training intervention).
  blood concentrations of eosinophils (EOSI) ) were collected (5 ml) in test tubes containing EDTA and analyzed using an automated cell counter (XN450; Sysmex, Norderstedt, Germany).
basophils | At baseline and at week 11(after the ten weeks of the training intervention).
  blood concentration of basophils (BASO) were collected (5 ml) in test tubes containing EDTA and analyzed using an automated cell counter (XN450; Sysmex, Norderstedt, Germany).

SECONDARY OUTCOMES:
Body composition | At baseline and after ten weeks of the training intervention.
  Body composition were determined, with barefoot and lightly dressed subjects, using a stadiometer (Holtain Ltd., UK) and an electronic scale (Tanita BC-533, Tokyo, Japan).
6 min walking test | At baseline and after ten weeks of the training intervention.
  The 6-minute walk test was performed before and after the training intervention as an indicator of exercise capacity.

CONTACTS AND LOCATIONS:
Locations (1):
- High Institute of Sports and Physical Education of Kef, Boulifa, Kef Governorate, Tunisia

IPD SHARING:
Plan to Share IPD: No
For confidentiality reasons, all data from this study are available upon request.